CLINICAL TRIAL: NCT04982601
Title: Evaluation of Yoga-Based Exercise Program for Females With Temporomandibular Disorders: A Randomized Clinical Trial
Brief Title: Yoga-Based Exercise Program For Temporomandibular Disorders
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medipol University (Other)
Responsible Party: Principal Investigator, ESRA ATILGAN, Associate Professor PhD, Medipol University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 10840098-07
Record Dates: First submitted 2021-07-08; First posted 2021-07-29 (Actual); Last update posted 2021-07-29 (Actual); Status verified 2021-07

CONDITIONS: Temporomandibular Disorders; Myofascial Pain Dysfunction Syndrome; Temporomandibular Joint Pain; Range of Motion; Yoga; Quality of Life
MeSH Terms: conditions — Temporomandibular Joint Disorders; Fibromyalgia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Yoga Group (Experimental): Yoga-based exercises were performed by a physiotherapist has Yoga training, by consisting of 10-person groups, 6 weeks, 3 days in a week for a total of 18 sessions. Yoga-based exercises are Hatha yoga-based sessions consisting of breathing exercises, warm-up exercises, relaxation, asanas exercises and lasts about one hour. Especially combined movements with upper extremity and neck movements and breathing exercises were used in breathing exercises. In the warm-up exercises, the muscles were extended by giving exercises especially for stretching the muscles. In this way, asanas were prepared. Asanas Ardra kati cahkrasana, padahastasana, trikosana, sasankasana, varaksana poses have been performed. Asanas were modified and applied according to the patient's condition. Relaxation exercises were used both after breathing exercises and at the end of the exercise program. With relaxation, the patients were allowed to leave their muscles relaxed with the whole body relaxation
  Interventions: Other: Yoga Exercises
- Control Group (No Intervention): No kind of intervention has been applied to control group they awaited for therapy procedure for 6 week. They have assessed at the end of the 6 weeks.

INTERVENTIONS:
Other: Yoga Exercises — Yoga-based exercises are Hatha yoga-based sessions consisting of breathing exercises, warm-up exercises, relaxation, asanas exercises.
  Arms: Yoga Group

SUMMARY:
Aims:The study was conducted to investigate the effect of Yoga-based exercise program on pain, range of motion(ROM), sleep quality, depression and quality of life in female patients with myofascial pain dysfunction(MPD) of temporomandibular disorders .

Methods: MPD will be included in the study. Yoga based exercise program will be performed to the first group as 3 times in a week for 6 weeks. The second group will be the control group. Outcome measurements; pain ,sleep quality, depression and quality of life will be evaluated. Evaluations will be repeated before and 6 weeks after exercise.

DETAILED DESCRIPTION:
Total 46 female patients between the ages of 20-50 planned to include in the study. In the study, 42 volunteers divided into two groups as yoga group (Group 1) and control group (Group 2). As a result of randomization, those chose 1 were taken in group 1, 2 were included in group 2. Yoga-based exercises performs for 6 weeks and 3 days in a week for the first group. The second group will be taken in the waiting list to be included in the program as a control group.

Yoga-based exercises perform by a physiotherapist has Yoga training, by consisting of 10-person groups, 6 weeks, 3 days in a week for a total of 18 sessions. Yoga-based exercises are Hatha yoga-based sessions consisting of breathing exercises, warm-up exercises, relaxation, asanas exercises and lasts about one hour.

Before the treatment, evaluations made immediately after the 6-weeks exercise program ended. As the primary outcome measures; jaw pain Visual Analog Scale (VAS), Neck Pain And Disability Scale (NPDS), neck and jaw range of motion (ROM) measurements; for secondary outcome measurements; the Pittsburg Sleep Quality Index (PUQI), Beck Depression Inventory (BDI) and Short Form 36 (SF36) are used. All measurements are repeated at the 6th week after yoga application and datas compared with the baseline measurements.

ELIGIBILITY:
Inclusion Criteria:

* Female patients aged 20-50 years diagnosed with MPD(myofascial pain dysfunction) syndrome according to the Research Diagnostic Criteria For Temporomandibular Disorders

Exclusion Criteria:

* Those with orthopedic problems such as degenerative arthritis and traumatic injuries, took physiotherapy program in the last 3 months and drug users were not included in the study.

Ages: 20 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — TMD has been reported that it is more common in women than men, as 5 times.
Enrollment: 39 (Actual)
Dates: Start 2014-01-07 (Actual); Primary Completion 2019-06-07 (Actual); Study Completion 2020-06-07 (Actual)

PRIMARY OUTCOMES:
Visual Analog Scale(VAS) | 6 weeks
  Pain intensity felt in the chin was evaluated with VAS at rest. They were asked to draw their pain level on a 10 cm scale between 0-10 points as 0=no pain, 10 unbearable pain
Neck Pain And Disability Scale (NPDS) | 6 weeks
  It is examined with Neck Pain and Disability Scale (NPDS). The severity of neck pain, duration of symptoms, and the disability of each item in the specified activities are evaluated. Each item is scored between 0-5 points. The total score is the sum of the points in each item and ranges from 0 to 100. High scores indicate more severe pain and effect
Neck and jaw range of motion (ROM) | 6 weeks
  The neck and chin area of the patients were measured with a ROM universal goniometer. While neck normal joint motion flexion (0-65 °), extension (50 °), lateral flexion (45 °) and rotation (60-80 °) were measured, TMJ movements, mandibular depression, protrusion, deviation movements were measured. Measurements were taken 3 times and the mean value was recorded

SECONDARY OUTCOMES:
Pittsburg Sleep Quality Index (PUQI) | 6 weeks
  Pittsburg Sleep Quality Index (PSQI) is a questionnaire that evaluates sleep quality with questions asked in 7 main topics as: subjective sleep quality, sleep latency, sleep duration, habitual sleep efficacy, sleep disorders, use of sleep medication and daytime functions. Questions are given a score between 0-3, high scores reflect poor sleep quality. Each of the seven main titles is evaluated first in itself. The scores of these components are added. Maximum 21 points are taken in total, and 5 points and above are considered as poor sleep quality
Beck Depression Inventory (BDI) | 6 weeks
  The depression level of the cases was evaluated using the Turkish version of the Beck Depression Inventory (BDI). Each of the items of the questionnaire examines somatic, affective and cognitive symptoms. Each item consists of 4 separate sentences that composed as showing increased severtiy about a specific symptom of depression. The sentences are scored between zero and three to indicate the severity of depression. High scores indicate more severe depression. The highest score that can be obtained in the survey is 63. For evaluation; 0-14 points shows mild depression, 15-29 points shows moderate depression, 30-63 points shows a serious depression level
Short Form 36 (SF36) | 6 weeks
  Turkish version of Short Form 36 (SF-36) was used to evaluate the quality of life. The SF-36 questionnaire with 36 items that measure eight health related quality of life domains: physical functioning (PF), social functioning (SF), role limitation due to physical problems (RP), role limitation due to emotional problems (RE), mental health (MH), energy and vitality (VT), bodily pain (BP), and general perception of health (GH). In the calculation of the results, each subscale is calculated separately. The scores of the subscales vary between 0 and 100, and the high score indicates good health

CONTACTS AND LOCATIONS:
Overall Officials: ESRA ATILGAN, PhD, Principal Investigator — Medipol University

IPD SHARING:
Plan to Share IPD: No